CLINICAL TRIAL: NCT00567047
Title: An Open-Label, Parallel-Group Study to Determine the Single and Multiple Dose Pharmacokinetics of Vildagliptin and Its Metabolites in Mild, Moderate or Severe Renal Impaired Patients Compared to Age, Sex and Weight-Matched Healthy Volunteers Following Daily Doses of 50 mg Vildagliptin for 14 Days
Brief Title: Pharmacokinetic Study of Vildagliptin in Patients With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237A2115
Record Dates: First submitted 2007-12-03; First posted 2007-12-04 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Type-2 Diabetes
MeSH Terms: interventions — Vildagliptin; 1-(((3-hydroxy-1-adamantyl)amino)acetyl)-2-cyanopyrrolidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Vildagliptin
  Interventions: Drug: vildagliptin

INTERVENTIONS:
Drug: vildagliptin
  Other Names: LAF237

SUMMARY:
This study will evaluate the pharmacokinetics of vildagliptin and its metabolites in patients with mild, moderate or severe renal impairment and healthy volunteers.

ELIGIBILITY:
Inclusion Criteria (general):

* Men and women (age 18 to 85 years)
* Participants must be nonfertile or using a medically approved birth control method. Additional information regarding this requirement available at screening
* Body mass index (BMI) ≤42 kg/m2 (inclusive)

Inclusion Criteria (for renal insufficient patients):

* Patients with mild, moderate, or severe kidney impairment. Please consult with participating physicians regarding the definitions of these levels of severity.
* Patients with diabetes must be treated with standard anti-diabetic therapy (diet and exercise, stable dose of sulfonylurea, insulin, or metiglinides) and agree to continue for the study duration

Inclusion Criteria (for healthy subjects):

* No current significant medical conditions as determined by history and physical.
* Serum creatinine with a calculated creatinine clearance (CrCl) of >80 ml/min.
* Matched to renal impaired patients in the study by age (±5 years), sex and weight (±10% BMI)
* Vital signs guided by the following ranges:

oral body temperature between 35.0-37.2 °C systolic blood pressure, 100-140 mm Hg diastolic blood pressure, 60-110 mm Hg pulse rate, 45-90 bpm

Exclusion criteria:

* Pregnant or lactating female.
* A history of type 1 diabetes, diabetes that is a result of pancreatic injury, or secondary forms of diabetes, acute metabolic diabetic complications (eg, ketoacidosis or hyperosmolar state (coma))
* Subjects that have been enrolled in previous vildagliptin studies or other DPP
* 4 inhibitor studies within six months
* History of renal transplant or immunosuppressant therapy
* Acute infections which may affect blood glucose control or other medical condition that may interfere with the interpretation of efficacy and safety data during the study
* Any pre-existing or history of diabetic ulcer
* Any of the following within the past 6 months: myocardial infarction (MI), coronary artery bypass surgery or percutaneous coronary intervention, unstable angina or stroke
* Any of the following electrocardiogram (ECG) abnormalities: Torsades de pointes, sustained and clinically relevant ventricular tachycardia or ventricular fibrillation, second degree atrioventricular (AV) block (Mobitz 1 and 2), third degree AV block, prolonged QTc (>500 ms)
* Malignancy including leukemia and lymphoma within the last 5 years.
* Liver disease such as cirrhosis or positive hepatitis B and C.
* Any alcohol related hepatic disease.
* Patients undergoing any method of dialysis
* Use of some concomitant medications
* Significant laboratory abnormalities as specified in the protocol
* History of active substance abuse (including alcohol) within the past 2 years.
* Smokers (i.e., 10 or more cigarettes per day)
* History of hypersensitivity to any of the study drugs or to drugs with similar chemical structures

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
• Pharmacokinetic measures | throughout the study

SECONDARY OUTCOMES:
• Safety and tolerability measures | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis investigative site
Locations (6):
- United States (5):
  - Novartis Investigator Site, Miami, Florida
  - Novartis Investigator Site, Orlando, Florida
  - Novartis Investigator Site, Minneapolis, Minnesota
  - Novartis Investigator Site, Knoxville, Tennessee
  - Novartis Investigator Site, Richmond, Virginia
- Novartis Investigator Site, Kiel, Germany